CLINICAL TRIAL: NCT02529917
Title: The Benefits of Hemp Protein Supplementation During Resistance Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Responsible Party: Principal Investigator, Phil Chilibeck, Ph.D., University of Saskatchewan
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 15-95
Record Dates: First submitted 2015-08-11; First posted 2015-08-20 (Estimated); Last update posted 2017-05-05 (Actual); Status verified 2017-05

CONDITIONS: Sarcopenia
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hemp powder (Experimental): Hemp powder supplement
  Interventions: Dietary Supplement: Hemp powder
- Soy powder (Active Comparator): Soy powder supplement
  Interventions: Dietary Supplement: Soy Powder

INTERVENTIONS:
Dietary Supplement: Hemp powder — Hemp powder supplement
  Arms: Hemp powder
Dietary Supplement: Soy Powder — Soy powder supplement
  Arms: Soy powder

SUMMARY:
Forty physically active men and women aged 18-45y will take part in an 8-week resistance training program, randomized (double blind) 1:1 into each of two groups. Twenty participants will be randomized to receive 60 g/d of hemp powder (containing approximately 40 g protein and 9 g oil) supplementation and 20 randomized to receive 60 g/d of soy supplementation (matched to the hemp for macronutrients and calories) during eight weeks of training. Each participant will complete testing before and after the intervention for assessment of body composition (lean tissue, fat, and bone mass), strength, central fatigue, markers of inflammation, and bone resorption. Over the 8-weeks of training, participants will train four-five days per week for 1-1.5 hours per session with exercises targeting all major muscle groups. The training will involve a "two day split" where different muscle groups are trained on two consecutive days (day 1 involves chest, back, and arms; day 2 legs, shoulders, and abdominals). Resistance training will provide the necessary stimulus for protein synthesis to optimize the effect of a protein-containing nutritional supplement. The hemp or soy powder will be consumed in two doses (i.e. 30 g powder containing 20 g protein per dose) immediately after exercise sessions and one hour after exercise. This dosing regimen is optimal for stimulating muscle protein synthesis and building muscle mass . On the one non-training day per week the two doses will be consumed with meals.

ELIGIBILITY:
Inclusion Criteria:

* At least 6 months experience with resistance training

Exclusion Criteria:

* Allergies to hemp or soy
* Consumption of other nutritional supplements in previous month
* Answered "yes" to questions on the Physical Activity Readiness Questionnaire

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2015-08; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change in lean tissue mass (kg) | 8 weeks
  Lean tissue mass measured with dual energy x-ray absrorptiometry

SECONDARY OUTCOMES:
Change in fat mass (kg) | 8 weeks
  Fat mass as measured by dual energy x-ray absorptiometry
Change in bone mass (grams) | 8 weeks
  Bone mass as measured by dual energy x-ray absorptiometry
Change in elbow flexor muscle thickness (cm) | 8 weeks
  Muscle thickness as assessed by ultrasound
Change in knee extensor muscle thickness (cm) | 8 weeks
  muscle thickness as measured by ultrasound
Change in bench press strength (kg) | 8 weeks
  Bench press strength as assess on a plate-loaded machine by the 1-RM method
Change in arm curl strength (kg) | 8 weeks
  Arm curl strength as assessed with dumbbells by the 1-RM method
Change in leg press strength (kg) | 8 weeks
  Leg press strength as assessed on a leg-press machine by the 1-RM method
Change in inflammation by interleukin-6 (mmol/l) levels | 8 weeks
  Interleukin-6 levels measured from saliva samples
Change in inflammation by C-reactive protein (mmol/l) levels | 8 weeks
  C-reactive protein levels measured from saliva samples
Change in bone resorption (N-telopeptides) (mmol/l) | 8 weeks
  N-telopeptides measured from urine samples
Change in voluntary muscle activation (Nm) | 8 weeks
  Voluntary muscle activation as measured by the interpolated twitch technique

CONTACTS AND LOCATIONS:
Overall Officials: Philip Chilibeck, Principal Investigator — University of Saskatchewan
Locations (1):
- University of Saskatchewan, Saskatoon, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kaviani M, Shaw KA, Candow DG, Farthing JP, Chilibeck PD. Effects of hemp supplementation during resistance training in trained young adults. Eur J Appl Physiol. 2024 Apr;124(4):1097-1107. doi: 10.1007/s00421-023-05337-7. Epub 2023 Oct 17. PMID 37847288